CLINICAL TRIAL: NCT02438917
Title: Biomarkers of Liver Fibrosis
Status: Terminated | Type: Observational
Why Stopped: collaborator Kinemend closed due to finances
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: KineMed (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 15-0548
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Cirrhosis; Biomarkers; Fibrosis
MeSH Terms: conditions — Hepatitis C; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Urine, Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hepatitis C: Patients who are about to begin HCV treatment

SUMMARY:
Chronic liver injury leads to the accumulation of proteins in the liver that form dense scars. Liver scar formation is typically a slow process that leads to major organ damage and loss of function over the course of many years. During scar formation the extracellular matrix in the liver changes. The type and quantity of extracellular collagen and other proteins change during tissue remodeling. Some of these changes can be detected by analyzing factors present in blood. Because of the lengthy time course, changes in the rate of liver scar formation and regression are very difficult measure; however, accurate measurements are needed in order to conduct trials of interventions aimed at preventing scar formation and/or promotion scar regression. Current methods have sub-optimal specificity and selectivity. The long term objective of the study is to identify serum proteins that can be used to accurately estimate rates of liver fibrosis progression and regression. The project focusses on a novel methodology that uses stable isotope labeling with deuterated water, D2O, to tag newly-synthesized proteins. Mass spectroscopy is used to identify individual proteins and to quantify the ratio of labeled protein to total protein. This ratio provides information about the rate of synthesis of the protein of interest. This method will be applied to specimens from patients with hepatitis C virus (HCV) infection who are about to begin HCV treatment. Treatment is known to reduce liver inflammation and collagen content.

DETAILED DESCRIPTION:
Chronic liver injury leads to the accumulation of proteins in the liver that form dense scars. Liver scar formation is typically a slow process that leads to major organ damage and loss of function over the course of many years. During scar formation the extracellular matrix in the liver changes. The type and quantity of extracellular collagen and other proteins change during tissue remodeling. Some of these changes can be detected by analyzing factors present in blood. Because of the lengthy time course, changes in the rate of liver scar formation and regression are very difficult measure; however, accurate measurements are needed in order to conduct trials of interventions aimed at preventing scar formation and/or promotion scar regression. Current methods have sub-optimal specificity and selectivity. The long term objective of the study is to identify serum proteins that can be used to accurately estimate rates of liver fibrosis progression and regression. The project focusses on a novel methodology that uses stable isotope labeling with deuterated water, D2O, to tag newly-synthesized proteins. Mass spectroscopy is used to identify individual proteins and to quantify the ratio of labeled protein to total protein. This ratio provides information about the rate of synthesis of the protein of interest. This method will be applied to specimens from patients with hepatitis C virus (HCV) infection who are about to begin HCV treatment. Treatment is known to reduce liver inflammation and collagen content.

The main questions being addressed are whether the regression of scar in the liver can be predicted based on the half-life of serum proteins and what is the identity of the proteins that are the best indicators of liver scar formation and regression.

The long term goal of the study is to develop a non-invasive test that can be used to estimate the extent of liver fibrosis and the rate of liver fibrosis generation and regression. Such a marker could be used to test drugs that promote fibrosis regression and/or prevent fibrogenesis and it could also be used to provide patients and healthcare providers with information about the extent of liver scarring.

Research is being done around the globe to determine develop innovative methods to accurately determine liver status. A metabolic labeling method will be tested in this project. This approach is based on the concept that liver status can be determined by measuring the ratio of newly-synthesized/pre-existing proteins. Patients will be given "heavy water" to drink. Heavy water contains D20. Deuterium is a stable isotope of hydrogen. Deuterium is not radioactive. It has been given to many patients and is considered to be entirely safe when administered according to the protocol that will be used in this study. Proteins that are synthesized during D20 labeling contain D20. Mass spectrometry is used to determine the percentages of scar proteins (and other indicator proteins) that are newly-synthesized. The analysis can be performed on a variety of tissues and bodily fluids. In this study, measurements will be made on blood, saliva, and urine samples from all the participants. Study subjects will be given the option of undergoing liver biopsy. The D20 content of biopsy tissue will be determined for the patients who elect this option.

The study group for this investigation is comprised of patients with chronic hepatitis C virus (HCV) infection who are about to begin HCV treatment. It is well established that HCV treatment reduces the amount of inflammation and scar in the liver. New treatments for HCV are far more effective and less toxic than earlier treatments. The treatment-induced changes in inflammation and hepatic scarring will impact the ratio of proteins in the metabolic labeling study. The rate of synthesis of scar proteins will go down and the ratio of new/pre-existing protein will change. Metabolic labeling data will be compared to other data about liver status, such as values of serum markers, liver stiffness measurements, and liver histopathology (when available).

Research will be performed at the Mount Sinai Medical Center, with coded, but de-identified specimens analyzed at Kinemed Patients initiating treatment for HCV infection are the source of potential subjects.

The final study group is expected to include 40 subjects. We expect about 2/3 of subjects who are approached to agree to participate and to sign the consent document. We expect 90% of the 40 subjects to complete the first 6 months of the study and we expect 80% to complete the entire study.

This is a single center study The duration of an individual subject's participation in the study: 36 months (including all follow up) The duration anticipated to enroll all study subjects: 6 months

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Positive test for HCV RNA
* Planning to initiate treatment for HCV in the near future
* Not diagnosed with any additional liver diseases, such as autoimmune hepatitis, hepatitis B, alcoholic liver disease, or HIV
* Able to travel to Mount Sinai
* Must understand and speak English
* Willing to sign informed consent and participate

Exclusion Criteria:

* Pregnancy
* Incarcerated Person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the hepatitis C virus (HCV) who are about to begin HCV treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Change in serum protein | baseline and 36 months
  Change in the ratio of transforming growth factor binding protein 1 (TGFB1) at 36 months as compared to baseline

SECONDARY OUTCOMES:
Change in the FibroScan score | baseline and 36 months
  Change in FibroScan score at 36 months as compared to baseline. FibroScan is performed to assess liver stiffness, an indicator of liver fibrosis.
Change in the ELF score | baseline and 36 months
  Change in ELF score at 36 months as compared to baseline
Change in the FIB-4 score | baseline and 36 months
  Change in the FIB-4 score at 36 months as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrea D Branch, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States